CLINICAL TRIAL: NCT01521091
Title: Comparison of Diagnostic Accuracy for Predicting Histology of Colorectal Lesions Using Magnifying Colonoscopy With Narrow Band Imaging, Indigo Carmine, and Acetic Acid Staining
Brief Title: Comparison of Diagnostic Accuracy for Predicting Histology of Colorectal Lesions
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjxhnk01
Record Dates: First submitted 2012-01-24; First posted 2012-01-30 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2012-01

CONDITIONS: Colorectal Neoplasms
Keywords: narrow band imaging（NBI）; indigo carmine; acetic acid; colorectal lesions; predicting histology
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All the lesions will be removed endoscopically or surgically and examine histologically by an independent gastrointestinal pathologist.
  Histological diagnosis is determined according to the World Health Organization (WHO) criteria. Pedunculated lesions are categorized according to Haggitt's classification.
Oversight: Data Monitoring Committee: No

SUMMARY:
Chromoendoscopy (indigo carmine or acetic acid) and Narrow Band Imaging (NBI) could make accurate evaluation in predicting of invasive depth of colorectal neoplasia. NBI could be the first choice.

DETAILED DESCRIPTION:
To compare the diagnostic accuracy of chromoendoscopy indigo carmine or acetic acid and NBI for differentiating neoplastic from non-neoplastic colorectal lesions, differentiating adenomas from carcinomas, and differentiating early carcinomas from invasive ones.

Included colorectal lesions consecutively distribute in a 1:1 ratio to 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with more than one lesion ≧ 6mm .

Exclusion Criteria:

* Patients with chronic inflammatory bowel disease, advanced cancer, insufficient bowel preparation, familial adenomatous polyposis (FAP)
* Lesions ≦ 5mm and submucosal tumor (SMT).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive adult patients undergoing colonoscopy and find out more than one lesion ≧ 6mm from Jan 2009 to Dec 2010.
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Li, MD. Ph.D, Principal Investigator — Departments of Gastroenterology and Clinical Laboratory, Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai,China,Shanghai Institute of Digestive Disease, Shanghai, China
Locations (1):
- Departments of Gastroenterology and Clinical Laboratory, Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China